CLINICAL TRIAL: NCT02600156
Title: A Pilot Study to Evaluate Magnetic Resonance Thermal Image-Guided Focal Laser Ablation of Prostate Cancer Tumors
Brief Title: Focal Laser Ablation of Low to Intermediate Prostate Cancer Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, David A. Woodrum, M.D., Ph.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-005500
Record Dates: First submitted 2015-09-04; First posted 2015-11-09 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Localized Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Experimental): MR guided focal laser ablation of prostate cancer using the Visualase Thermal Therapy System.
  Interventions: Procedure: Focal laser ablation of the prostate

INTERVENTIONS:
Procedure: Focal laser ablation of the prostate — MR guided laser ablation of the focal prostatic lesion which has been identified by MRI and biopsy prior to ablation.
  Other Names: Visualase Laser Ablation

SUMMARY:
The primary purpose of this study is to evaluate the feasibility and safety of MRI-guided focal laser ablation (Laser-Induced Interstitial Thermal Therapy, LITT) to treat low-risk native prostate cancer.

DETAILED DESCRIPTION:
The study is being done to evaluate the safety and effectiveness of Magnetic Resonance Imaging (MRI)-guided focal laser therapy with the Visualase Thermal Therapy System to treat low-risk prostate cancer tumors. Unlike surgery or radiotherapy which affects a large portion of the prostate or the entire organ, localized or focal therapy is intended to treat a small portion of tissue in which the cancer has been found by biopsy.

ELIGIBILITY:
Inclusion Criteria

* Male, 45 years of age or older.
* Diagnosis of prostate adenocarcinoma.
* Clinical stage T1c or T2a.
* Gleason score of 7 (3+4 or 4+3) or Intermediate risk Gleason 6
* PSA less than or equal to 20 ng/mL
* Three or fewer biopsy locations with prostate cancer which correlate with MRI findings.
* No lesion > or = 2cm
* One, two, or three tumor suspicious regions identified on multiparametric MRI
* No definite radiographic indication of extra-capsular extension.
* Estimated survival of 5 years or greater, as determined by treating physician.
* Tolerance for anesthesia/sedation.
* Ability to give informed consent.

Exclusion Criteria

* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI.
* History of other primary non-skin malignancy within previous three years.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Success rate | 3 years
  To evaluate the procedural success rate of using the MR-guided laser ablation to target, access, thermally monitor, and focally ablate MR-visible prostate cancer lesions.
Incidence of treatment emergent adverse events | 3 years
  To evaluate patient-related safety by monitoring short and long-term complications related to the procedure such as but not limited to incontinence, impotence, and urethral fistulas.

SECONDARY OUTCOMES:
Short- and mid-term ablative success | 3 years
  To obtain preliminary data on ablative success using longitudinal MR imaging assessment of treated areas.

CONTACTS AND LOCATIONS:
Overall Officials: David Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials